CLINICAL TRIAL: NCT06746844
Title: A Comparative Study Between ViewMind AtlasTM, a Novel Digital Measure of Cognition, and Traditional Cognitive Tests
Brief Title: ViewMind Atlas Cognition
Acronym: VM-Cog
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: ViewMind (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ViewMindRM
Record Dates: First submitted 2024-11-29; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-07

CONDITIONS: MCI; Cognitive Ability, General; Cognitive Decline; Cognition
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cognitive assessment group (Experimental): All participants will undergo cognitive evaluation using VM Atlas and traditional tests
  Interventions: Device: ViewMind Atlas™

INTERVENTIONS:
Device: ViewMind Atlas™ — The intervention involves the use of ViewMind Atlas™, a novel digital tool for cognitive assessment, and traditional cognitive tests. The ViewMind Atlas™ device evaluates cognitive performance through eye-tracking technology and advanced analytics, providing objective measurements of cognitive function. Traditional cognitive tests are used as the standard comparator to validate the device's diagnostic performance

SUMMARY:
The objective of this study is to demonstrate the clinical validity, analytical validity and safety of ViewMind Atlas as an adjunctive tool to be used by healthcare professionals (HCP) evaluating cognitive impairment in adults aged 45 to 95 years old.

DETAILED DESCRIPTION:
This will be a comparative study in which each subject undergoes testing by certified HCP evaluators administering the and ViewMind AtlasTM evaluation and the MoCA test, as well as additional tests, which are part of a reference standard neurocognitive battery of tests for cognition (WAT-BA, BEM-144, Rey Complex Figure Test, Wechsler Memory Scale subtests, WAIS III subtests, Trail Making Test A and B, Boston Naming Test, Phonological Verbal Fluency test, Semantic Verbal Fluency test, and Clock Drawing Test). Test-retest reliability of ViewMind AtlasTM will be conducted one week after initial testing.

Primary Objective:

● To assess the clinical validity of ViewMind Atlas for identifying cognitive impairment, as determined by MoCA

Secondary Objectives:

* To demonstrate the analytical validity of ViewMind Atlas for measuring cognition (evaluated) against an appropriate reference standard (MoCA)
* To examine the discriminant and convergence validity between ViewMind AtlasTM and a battery of neurocognitive tests in identifying cognitively healthy and cognitively impaired test subjects.
* To compare the test-retest reliability of ViewMind AtlasTM.
* To assess the safety of the ViewMind system.

  1. Sensitivity (Se), Specificity (Sp) Negative Predictive Value (NPV), Positive Predictive Value (PPV) positive likelihood ratios, and negative likelihood ratios and Accuracy of ViewMind AtlasTM agreement with the classification of MoCA in identifying cognitively healthy and cognitively impaired test participants.
  2. Correlation between the results obtained with ViewMind Atlas™ and the scores of each component of the MoCA test
  3. Correlation between the results obtained with ViewMind Atlas™ and the scores of each component of the neurocognitive test battery
  4. Regression analysis of test-retest reliability for ViewMind AtlasTM.
  5. Collection of adverse events (AEs) Total no. of subjects: 327
* n= 128 for test-retest of ViewMind This study will be conducted in one site: Ramos Mejia Hospital, in Buenos Aires, Argentina.

This study is estimated to last 16 weeks, from start of enrollment to final data analysis.

All participants will attend at least a single visit during which the cognitive evaluations will be carried out. 128 participants will then come back for a second visit 1-3 weeks after the first visit, to undergo another cognitive evaluation with ViewMind.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Male or female, aged between 45 and 95 years.
* Cohort 1: Presence of cognitive complaints and objectively measured cognitive impairment of an MMSE of > 26, such as memory loss or other cognitive difficulties (60% of the overall study population). These complaints can be self-reported or noted by a close family member. Diagnosis of MCI by PI or delegated qualified provider on the study team.
* Cohort 2: Absence of cognitive complaints and absence of objectively measured cognitive impairment as determined by MMSE > 26 and neuropsychological tests. Diagnosis of CN by PI or delegated qualified provider on the study team (40% of the overall study population).
* Willing to sign written informed consent and ability to comply with study requirements.
* Have adequate vision and hearing, with or without corrective devices, to ensure accurate self-reporting and comprehension of study materials.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Participants with dementia, defined here as an MMSE of < 25 and diagnosis of cognitive decline that is not MCI but more severe in nature by the PI or delegated qualified provider on the study team.
* Advanced, severe progressive or unstable disease that may interfere with the safety, tolerability and study assessments, or put the participant at special risk as judged by the investigator.
* Subjects who had received an investigational drug or therapy within 30 days or 5 half-lives, whichever was longer, of the first visit.
* Participants with glaucoma, cataract, macular degeneration in both eyes, or any other cause of uncorrected visual impairment (less than 20/30).
* Participants with severe color-blindness.
* Participants with developmental cognitive dysfunction (congenital, pediatric).
* Major psychiatric disorder (e.g., chronic psychosis, recurrent depressive disorder, generalized anxiety disorder).
* Use of cognitive enhancing drugs (e.g., cholinesterase inhibitors).
* A concurrent diagnosis of epilepsy.
* History of alcohol misuse and/or illicit drug use.
* History of acute damage, including stroke, traumatic brain injury, tumors, etc.
* Presence of sleep apnea.
* Recent participation in another neuropsychological study.

Ages: 45 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2024-12-16 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of ViewMind Atlas™ in Identifying Cognitive Impairment | At baseline (Visit 1)
  Evaluate the sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), accuracy, and likelihood ratios (positive and negative) of ViewMind Atlas™ compared to clinical diagnosis rendered by qualified providers using standard neuropsychological assessments.

CONTACTS AND LOCATIONS:
Overall Officials: María B Eizaguirre, PhD, Study Chair — Multiple Sclerosis University Center, Ramos Mejía Hospital, Buenos Aires, Argentina.
Locations (1):
- Ramos Mejía Hospital, Buenos Aires City, Buenos Aires, Argentina